CLINICAL TRIAL: NCT07113574
Title: Pharmacokinetics of Meropenem and Aztreonam After Intraperitoneal Administration Via Cycler-therapy in APD Patients Without Peritonitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karl Landsteiner Insitute for Nephrology and Haemato-Oncology (Network)
Collaborators: Karl Landsteiner University of Health Sciences (Other); Medical University of Cologne (Other); University Hospital St. Polten (Other); University of Vienna (Other)
Responsible Party: Principal Investigator, Dominik Tüchler, MD, Karl Landsteiner Insitute for Nephrology and Haemato-Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS1-EK-2/483-2020
Record Dates: First submitted 2025-07-10; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Peritoneal Dialysis Associated Peritonitis; Peritoneal Dialysis (PD); Peritoneal Dialysis; Peritoneal Dialysis, Continuous Ambulatory; Meropenem; Aztreonam; Antibacterial Agents; Intraperitoneal Antibiotics; Kidney Failure, Chronic; Anti-Bacterial Agents; Drug Therapy
Keywords: Pharmacokinetics; meropenem; aztreonam; intraperitoneal administration; automated cycler-therapy; APD patients; peritonitis
MeSH Terms: conditions — Kidney Failure, Chronic; Peritonitis | interventions — Meropenem; Aztreonam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraperitoneal meropenem via cycler-therapy in APD (Experimental): Intraperitoneal administration of meropenem via cycler-therapy in automated peritoneal dialysis patients without peritonitis
  Interventions: Drug: Meropenem 1000 mg; Other: automated peritoneal dialysis with following long time dwell; Diagnostic Test: Sampling
- intraperitoneal aztreonam via cycler-therapy in APD (Experimental): Intraperitoneal administration of aztreonam via cycler-therapy in automated peritoneal dialysis patients without peritonitis
  Interventions: Drug: Aztreonam 2000 mg; Other: automated peritoneal dialysis with following long time dwell; Diagnostic Test: Sampling

INTERVENTIONS:
Drug: Meropenem 1000 mg — Administration of meropenem after intraperitoneal administration via cycler-therapy in APD patients without peritonitis
  Arms: intraperitoneal meropenem via cycler-therapy in APD
Drug: Aztreonam 2000 mg — Administration of aztreonam after intraperitoneal administration via cycler-therapy in APD patients without peritonitis
  Arms: intraperitoneal aztreonam via cycler-therapy in APD
Other: automated peritoneal dialysis with following long time dwell — The cycler therapy, followed by a prolonged dwell, will be performed as outlined in the study protocol.
Diagnostic Test: Sampling — The sampling of blood, dialysate, and urine will be performed as outlined in the study protocol.

SUMMARY:
Peritoneal dialysis-associated peritonitis (PDAP) remains one of the most serious complications in patients undergoing peritoneal dialysis (PD), contributing significantly to hospitalization, technique failure, and mortality. Intraperitoneal (IP) antibiotic administration is the standard of care in PDAP, as it provides high local drug concentrations at the site of infection. However, dosing recommendations are largely based on pharmacokinetic (PK) studies in continuous ambulatory peritoneal dialysis (CAPD) patients. Automated peritoneal dialysis (APD), now widely used, differs significantly from CAPD in terms of dialysate volumes, frequency of exchanges, and peritoneal clearance. As a result, extrapolation of CAPD-based dosing regimens may lead to antibiotic underdosing in APD patients.

This prospective, open-label, single-center descriptive PK study investigates the plasma and dialysate concentration-time profiles of meropenem and aztreonam after IP administration into the short-dwell cycler exchanges during nighttime APD. The rationale is that administration into the early short dwells may ensure adequate antibiotic levels both during active cycling (when frequent exchanges may clear the drug rapidly) and during the subsequent long daytime dwell through back-diffusion from systemic circulation.

Twelve stable APD patients without peritonitis will be enrolled (6 per drug group). Inclusion requires patients to be on a stable APD regimen for at least one month using glucose-based dialysate for short nighttime dwells and Icodextrin for the daytime dwell. Patients with current infections, recent peritonitis, or significant comorbid conditions are excluded.

On the study day, each participant will receive either:

Meropenem: 0.75 g added to a 5L glucose-based peritoneal dialysis fluid (PDF) bag, or

Aztreonam: 2 g prepared similarly.

The antibiotic-containing 5L PDF bag is used as the first bag in the APD cycler session, followed by a second 5L antibiotic-free PDF bag, yielding a total of five 2L nighttime exchanges. After cycler therapy, a 1.5L Icodextrin fill is instilled for the long daytime dwell.

Sampling includes:

Venous blood: at 0 (pre-dose), 1, 2, 4.5, 6.5, 9, 10, 12, 16, and 24 hours.

Dialysate: inflow/outflow from each cycle and at defined intervals during the Icodextrin dwell (up to 24 hours).

Urine: 5 mL from a 24-hour collection in patients with residual renal function.

Drug concentrations in plasma, dialysate, and urine will be quantified using validated high-performance liquid chromatography (HPLC) techniques. Primary PK endpoints include area under the curve (AUC), maximum plasma concentration (Cmax), time to reach Cmax (Tmax), and half-life (t½) in each compartment. Secondary endpoints include ratios of AUC and Cmax across compartments, time above the minimal inhibitory concentration (T>MIC), and AUC0-24/MIC.

This study does not include formal hypothesis testing but aims to generate descriptive PK data to inform optimized dosing of meropenem and aztreonam for APD patients. Currently, there is a lack of pharmacokinetic data guiding IP antibiotic dosing specifically in APD. The study's findings may support more accurate and effective antibiotic administration protocols for PDAP and potentially for the treatment of other systemic infections (e.g., pneumonia) in this population.

The anticipated benefit is improved antimicrobial efficacy through better PK/PD target attainment while avoiding the need for intravenous therapy. The risk to participants is minimal, consisting primarily of standard procedures (blood draws, single-dose IP drug administration). Ethical approval has been obtained, and all participants will provide written informed consent. The study complies with Good Clinical Practice (GCP) and relevant regulatory and ethical standards, including the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged over 18 years
* Patients on a stable APD regime for at least 1 month
* Patients on an APD regime using a glucose-based PDF (1,36% and/or 2,27%) for short nighttime dwells and Icodextrin for the long daytime dwell
* Willingness and ability to comply with the protocol
* Signed informed consent

Exclusion Criteria:

* Any systemic infection
* Peritonitis or catheter-related infection which required antibiotic treatment within 2 months prior to the start of the study
* Allergy or hypersensitivity against study drug
* Severe hepatic impairment (Child-Pugh Class C)
* Pregnancy, or women of childbearing potential not willing to apply adequate contraception during study period
* Any disease considered relevant for proper performance of the study or risks to the patient, at the discretion of the investigator
* Hemoglobin below 9 g/dl
* BMI below 19 or above 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | 24 hours
Maximum concentration (Cmax) | 24 hours
Time to Cmax (Tmax) | 24 hours
Half-life (t½) | 24 hours

SECONDARY OUTCOMES:
Time above minimum inhibitory concentration (T>MIC) | 24 hours
AUC0-24/MIC | 24 hours
Compartmental ratios (AUC, Cmax) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martin F Wiesholzer, MD, Principal Investigator — UK St. Pölten
Locations (1):
- UK St. Pölten, Sankt Pölten, Austria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] de Vin F, Rutherford P, Faict D. Intraperitoneal administration of drugs in peritoneal dialysis patients: a review of compatibility and guidance for clinical use. Perit Dial Int. 2009 Jan-Feb;29(1):5-15. PMID 19164246
- [Background] Kussmann M, Schuster L, Wrenger S, Pichler P, Reznicek G, Burgmann H, Poeppl W, Zeitlinger M, Wiesholzer M. Influence of Different Peritoneal Dialysis Fluids on the In Vitro Activity of Cefepime, Ciprofloxacin, Ertapenem, Meropenem and Tobramycin Against Escherichia Coli. Perit Dial Int. 2016 11-12;36(6):662-668. doi: 10.3747/pdi.2015.00161. Epub 2016 Sep 28. PMID 27680756
- [Background] Wiesholzer M, Pichler P, Reznicek G, Wimmer M, Kussmann M, Balcke P, Burgmann H, Zeitlinger M, Poeppl W. An Open, Randomized, Single-Center, Crossover Pharmacokinetic Study of Meropenem after Intraperitoneal and Intravenous Administration in Patients Receiving Automated Peritoneal Dialysis. Antimicrob Agents Chemother. 2016 Apr 22;60(5):2790-7. doi: 10.1128/AAC.02664-15. Print 2016 May. PMID 26902765
- [Background] Warady BA, Bakkaloglu S, Newland J, Cantwell M, Verrina E, Neu A, Chadha V, Yap HK, Schaefer F. Consensus guidelines for the prevention and treatment of catheter-related infections and peritonitis in pediatric patients receiving peritoneal dialysis: 2012 update. Perit Dial Int. 2012 Jun;32 Suppl 2(Suppl 2):S32-86. doi: 10.3747/pdi.2011.00091. No abstract available. PMID 22851742
- [Background] Peerapornratana S, Chariyavilaskul P, Kanjanabuch T, Praditpornsilpa K, Eiam-Ong S, Katavetin P. Short-Dwell Cycling Intraperitoneal Cefazolin Plus Ceftazidime in Peritoneal Dialysis Patients. Perit Dial Int. 2017 Mar-Apr;37(2):218-224. doi: 10.3747/pdi.2015.00300. Epub 2016 Oct 13. PMID 27738089
- [Background] Manley HJ, Bailie GR. Treatment of peritonitis in APD: pharmacokinetic principles. Semin Dial. 2002 Nov-Dec;15(6):418-21. doi: 10.1046/j.1525-139x.2002.00103.x. PMID 12437537
- [Background] Salzer W. Antimicrobial-resistant gram-positive bacteria in PD peritonitis and the newer antibiotics used to treat them. Perit Dial Int. 2005 Jul-Aug;25(4):313-9. PMID 16022084
- [Background] Van Ende C, Tintillier M, Cuvelier C, Migali G, Pochet JM. Intraperitoneal meropenem administration: a possible alternative to the intravenous route. Perit Dial Int. 2010 Mar-Apr;30(2):250-1. doi: 10.3747/pdi.2009.00052. No abstract available. PMID 20200373
- [Background] Li PK, Szeto CC, Piraino B, de Arteaga J, Fan S, Figueiredo AE, Fish DN, Goffin E, Kim YL, Salzer W, Struijk DG, Teitelbaum I, Johnson DW. ISPD Peritonitis Recommendations: 2016 Update on Prevention and Treatment. Perit Dial Int. 2016 Sep 10;36(5):481-508. doi: 10.3747/pdi.2016.00078. Epub 2016 Jun 9. No abstract available. PMID 27282851
- [Background] Hsieh YP, Chang CC, Wang SC, Wen YK, Chiu PF, Yang Y. Predictors for and impact of high peritonitis rate in Taiwanese continuous ambulatory peritoneal dialysis patients. Int Urol Nephrol. 2015 Jan;47(1):183-9. doi: 10.1007/s11255-014-0763-5. Epub 2014 Jul 18. PMID 25034275
- [Background] Szeto CC, Wong TY, Chow KM, Leung CB, Li PK. Are peritoneal dialysis patients with and without residual renal function equivalent for survival study? Insight from a retrospective review of the cause of death. Nephrol Dial Transplant. 2003 May;18(5):977-82. doi: 10.1093/ndt/gfg027. PMID 12686674
- [Background] Perez Fontan M, Rodriguez-Carmona A, Garcia-Naveiro R, Rosales M, Villaverde P, Valdes F. Peritonitis-related mortality in patients undergoing chronic peritoneal dialysis. Perit Dial Int. 2005 May-Jun;25(3):274-84. PMID 15981776
- [Background] Ghali JR, Bannister KM, Brown FG, Rosman JB, Wiggins KJ, Johnson DW, McDonald SP. Microbiology and outcomes of peritonitis in Australian peritoneal dialysis patients. Perit Dial Int. 2011 Nov-Dec;31(6):651-62. doi: 10.3747/pdi.2010.00131. Epub 2011 Jun 30. PMID 21719685
- [Background] Davenport A. Peritonitis remains the major clinical complication of peritoneal dialysis: the London, UK, peritonitis audit 2002-2003. Perit Dial Int. 2009 May-Jun;29(3):297-302. PMID 19458302
- [Background] Brown MC, Simpson K, Kerssens JJ, Mactier RA; Scottish Renal Registry. Peritoneal dialysis-associated peritonitis rates and outcomes in a national cohort are not improving in the post-millennium (2000-2007). Perit Dial Int. 2011 Nov-Dec;31(6):639-50. doi: 10.3747/pdi.2010.00185. Epub 2011 Jul 31. PMID 21804138
- [Background] Boudville N, Kemp A, Clayton P, Lim W, Badve SV, Hawley CM, McDonald SP, Wiggins KJ, Bannister KM, Brown FG, Johnson DW. Recent peritonitis associates with mortality among patients treated with peritoneal dialysis. J Am Soc Nephrol. 2012 Aug;23(8):1398-405. doi: 10.1681/ASN.2011121135. Epub 2012 May 24. PMID 22626818